CLINICAL TRIAL: NCT05770791
Title: Comparative Effects of Using Black Seed (Nigella Sativa) and Cumin Seed ( Cuminum Cyminum) on Body Composition Profile of Obese Grade I
Brief Title: Comparative Effects of Using Black Seed and Cumin Seed on BCP of Obese Grade I
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sehat Medical Complex (Other)
Responsible Party: Principal Investigator, Waseem Javaid, Project Director, Sehat Medical Complex
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ZaraYameen001-23
Record Dates: First submitted 2023-02-19; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-02

CONDITIONS: Obese
Keywords: Cumin Seeds; Black seed; Obese grade I
MeSH Terms: conditions — Obesity | interventions — Nigella sativa oil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A Obese Grade I
  Interventions: Dietary Supplement: Black Seed ( Nigella Sativa)
- Group B (Active Comparator): Group B Obese Grade I
  Interventions: Dietary Supplement: Cumin Seed (Cuminum Cyminum)

INTERVENTIONS:
Dietary Supplement: Black Seed ( Nigella Sativa) — Intervention will be given once a day for 1 month, total 30 days Data will be collected at baseline and at the end of the intervention at 30th day
  Arms: Group A
Dietary Supplement: Cumin Seed (Cuminum Cyminum) — Intervention will be given once a day for 1 month, total 30 days Data will be collected at baseline and at the end of the intervention at 30th day
  Arms: Group B

SUMMARY:
The goal of this Randomized clinical trial is to compare effectiveness of of using black seed (Nigella sativa) and cumin seed (Cuminum cyminum) on Body composition profile of obese grade 1. The primary objective of this study is To compare effectiveness of of using black seed (Nigella sativa) and cumin seed (Cuminum cyminum) on Body composition profile of obese grade 1. Subjects will be given a consent form and after subjects read and sign the informed consent, they would be included in study according to eligibility criteria.

DETAILED DESCRIPTION:
Obesity is a global pandemic that is associated with high morbidity and mortality. Natural herbs are commonly used for weight reduction and appetite suppression. Worldwide data based on 1698 studies has shown that the global prevalence of obesity has increased from 3.2 to 10.8% in men and from 6.4 to 14.9% in women. Meanwhile, herbal products are marketed for their weight-loss properties, such as Nigella sativa which has been used for centuries to treat rheumatoid arthritis, diabetes, and asthma; recently, the anti-obesity characteristics of N. sativa have also been indicated. The antihyperglycemic activity, inhibition of free radical formation, anti-obesity and anti-inflammatory activity of cumin seed extract have also been reported previously.

ELIGIBILITY:
Inclusion Criteria:

* Subject having BMI between 30 kg/m2 - 34.5 kg/m2

Exclusion Criteria:

* Subjects having kidney or liver problems
* Having ulcers in GIT
* Subjects having hypertension, thyroid, diabetes or cardiovascular disorders
* Pregnant and lactating mothers
* Subjects who are using hormonal or anti-obesity medications

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-01-27 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Body Composition Profile | Change from baseline at 30th Day
  permits a detailed analysis of the body's major structural components like muscle mass, fat, and bone. It is measured in percentage.

SECONDARY OUTCOMES:
BMI | Change from Baseline at 30th Day
  Body mass index is a value derived from the mass and height of a person. The BMI is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m², resulting from mass in kilograms and height in metres

CONTACTS AND LOCATIONS:
Overall Officials: Momina Mehmood, Principal Investigator — University of Lahore
Locations (1):
- Sehat Medical Complex, Lahore, Lahore, Punjab Province, Pakistan